CLINICAL TRIAL: NCT00120692
Title: An Open-Label, Randomized Phase 2 Study to Validate a Patient Satisfaction Questionnaire for Anemia Treatment in Female Breast Cancer Patients Treated With Darbepoetin Alfa or Recombinant Human Erythropoietin for Anemia Due to Chemotherapy
Brief Title: Treatment for Patients Suffering From Anemia Due to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020152
Record Dates: First submitted 2005-06-30; First posted 2005-07-19 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer; Anemia
Keywords: breast cancer; darbepoetin alfa; Amgen
MeSH Terms: conditions — Breast Neoplasms; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa
Drug: Recombinant Human Erythropoietin

SUMMARY:
The purpose of this study is to validate a Patient Satisfaction Questionnaire for Anemia Treatment (PSQ-AT) in female breast cancer patients treated with darbepoetin alfa or recombinant human erythropoietin (rHuEPO) for anemia due to chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Female subjects receiving multi-cycle chemotherapy - Anemia due to chemotherapy (hgb less than or equal to 11.0 g/dL) - Expected to receive greater than or equal to 8 additional weeks of chemotherapy as part of their planned treatment - Karnofsky Performance Scale (KPS) greater than or equal to 50% - Adequate renal function - Adequate liver function Exclusion Criteria: - Iron deficiency - Unstable cardiac disease - Known positive test for human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Anemia correction

SECONDARY OUTCOMES:
Activities of daily living, patient preference

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Senecal FM, Yee L, Gabrail N, Charu V, Tomita D, Rossi G, Schwartzberg L. Treatment of chemotherapy-induced anemia in breast cancer: results of a randomized controlled trial of darbepoetin alfa 200 microg every 2 weeks versus epoetin alfa 40,000 U weekly. Clin Breast Cancer. 2005 Dec;6(5):446-54. doi: 10.3816/cbc.2005.n.050. PMID 16381629
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com